CLINICAL TRIAL: NCT02043223
Title: Stopping Postpartum Vitamin A Supplementation: Are we Missing Concealed Benefit?
Brief Title: Stopping Postpartum Vitamin A Supplementation: Missing Concealed Benefit
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Peter Bergman, MD, PhD (Unknown); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-13060
Record Dates: First submitted 2013-12-05; First posted 2014-01-23 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Vitamin A Deficiency
Keywords: Vitamin A; Breast milk; Postpartum vitamin A supplementation; Infant vaccine response
MeSH Terms: conditions — Vitamin A Deficiency | interventions — Vitamin A; Postpartum Period

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Early postpartum vitamin A suppl. (Experimental): Single dose 200,000 IU vitamin A supplementation at <3-day and placebo supplementation at 6-wk postpartum.
  Interventions: Dietary Supplement: Vitamin A (<3-day postpartum)
- Late postpartum vitamin A suppl. (Experimental): Placebo supplementation at <3-day and single dose 200,000 IU vitamin A supplementation at 6-wk postpartum.
  Interventions: Dietary Supplement: Vitamin A (6 wk postpartum)
- Early & late postpartum vitamin A suppl (Experimental): 200,000 IU vitamin A supplementation, both at <3-day and 6-wk postpartum
  Interventions: Dietary Supplement: Vitamin A (<3-day and 6 wk postpartum)
- No postpartum vitamin A suppl. (Experimental): Placebo supplementation, both at <3-day and 6-wk postpartum.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A (<3-day postpartum) — Single dose 200,000 IU vitamin A supplementation at <3-day and placebo supplementation at 6-wk postpartum.
  Arms: Early postpartum vitamin A suppl.
Dietary Supplement: Vitamin A (6 wk postpartum) — Placebo supplementation at <3-day and single dose 200,000 IU vitamin A supplementation at 6-wk postpartum.
  Arms: Late postpartum vitamin A suppl.
Dietary Supplement: Vitamin A (<3-day and 6 wk postpartum) — 200,000 IU vitamin A supplementation, both at <3-day and 6-wk postpartum
  Arms: Early & late postpartum vitamin A suppl
Dietary Supplement: Placebo — Placebo supplementation, both at <3-day and 6-wk postpartum.
  Arms: No postpartum vitamin A suppl.

SUMMARY:
The purpose of this study is to evaluate the effect of post-partum maternal vitamin A supplementation on breast milk bioactive compounds and immune status, growth and morbidity of children in the first four months of life.

DETAILED DESCRIPTION:
The effect will be assessed by the milk and blood.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women >-18 years of age with low-risk obstetric

Exclusion Criteria:

* Pregnant women expecting a multiple birth
* Take vitamin A supplements during postpartum apart from study intervention
* Premature birth
* Newborn babies with birth defects and / or other serious diseases

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Breast milk immune regulators | Four months
  immune regulators in breast milk e.g. B-cell activating factor (BAFF); IL-7; Lactoferrin; sCD14, sIgA and TGF-beta levels at three time points-
  1. < 3-day postpartum (before 1st dose of supplementation)
  2. 7 wk postpartum (1wk after 2nd dose of supplementation)
  3. 15 wk postpartum

SECONDARY OUTCOMES:
Infant T helper cell immune responses | Four months
  Mitogen stimulated whole blood IL-10, IL-13, IFN-gamma, IL-21 and IL-17 responses at two time points-
  1. 7 wk of age (1wk after 2nd dose of maternal supplementation , as well as, 1wk after first doses of pentavalent vaccination)
  2. 15 wk of age (1wk after three doses of pentavalent vaccination)
Infant innate immune responses | Four months
  Tall like receptor (TLR)-4 and TLR9 agonist stimulated whole blood TNF-alpha and IL-10 and IFN-alpha responses at two time points-
  1. 7 wk of age (1wk after 2nd dose of maternal supplementation , as well as, 1wk after first doses of pentavalent vaccination)
  2. 15 wk of age (1wk after three doses of pentavalent vaccination)
Infant vaccines (Hepatitis B, Tetanus and Oral polio) specific antibody responses | Four months
  Hepatitis B and Tetanus Toxoid specific plasma cell IgG responses at 15 wk of age (1wk after three doses of pentavalent vaccination) And Hepatitis B and Tetanus Toxoid specific IgG in plasma and Polio (3 serotypes) specific secretory IgA (sIgA) in stool at two time points-
  1. 7 wk of age (1wk after 2nd dose of maternal supplementation , as well as, 1wk after first doses of pentavalent vaccination)
  2. 15 wk of age (1wk after three doses of pentavalent vaccination)
Relative abundance of infant gut microbial community and gut inflammatory markers | Four months
  Next generation sequencing (NGS) of bacterial 16s rDNA (+qPCR) in extracted stool samples and assessment of infant gut inflammatory markers e.g. human β-defensin-2 (HBD2); Neopterin; α-1-antitrypsin (AAT); neutrophil gelatinase-associated lipocalin (NGAL)-2 and S100A at two time points-
  1. 7 wk of age (1wk after 2nd dose of maternal supplementation , as well as, 1wk after first doses of pentavalent vaccination)
  2. 15 wk of age (1wk after three doses of pentavalent vaccination)

OTHER OUTCOMES:
Infant vitamin A status | Four months
  Infant plasma vitamin A status at 7 wk and 15 wk of age
Infant growth | Four months
  Infant Weight-for-Age z-score (WAZ) at 7 wk and 15 wk of age
Infant morbidity | Four months
  Infant morbidity status up to four months of age
Mother vitamin A status | Four months
  Plasma Retinol Binding Protein (RBP) and breast milk vitamin A level at two time points-
  1. < 3-day postpartum (before 1st dose of supplementation)
  2. 15 wk postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Shaikh M Ahmad, Ph.D, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Ahmad SM, Hossain MI, Bergman P, Kabir Y, Raqib R. The effect of postpartum vitamin A supplementation on breast milk immune regulators and infant immune functions: study protocol of a randomized, controlled trial. Trials. 2015 Mar 31;16:129. doi: 10.1186/s13063-015-0654-9. PMID 25872802